CLINICAL TRIAL: NCT01093924
Title: Partnerships to Overcome Obesity Disparities in Hawaii
Brief Title: Partnerships to Overcome Obesity Disparities in Hawaii: 18-month CBPR Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PILI 'Ohana 5 year; R24MD001660-04 (NIH)
Record Dates: First submitted 2010-03-17; First posted 2010-03-26 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Obesity
Keywords: Behavioral weight loss maintenance intervention; Weight loss; Weight loss maintenance
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- self-guided weight loss maintenance (No Intervention): 15-month self-guided weight loss maintenance group will receive monthly reminders to maintain their weight loss and newsletters that contain health information.
- DVD group (Experimental): 15-month weight loss maintenance intervention deliver via DVD.
  Interventions: Behavioral: PILI 'Ohana 18-month weight loss maintenance
- face-to-face group (Experimental): 15-month weight loss/weight loss maintenance intervention delivered in a group setting
  Interventions: Behavioral: PILI 'Ohana 18-month weight loss maintenance

INTERVENTIONS:
Behavioral: PILI 'Ohana 18-month weight loss maintenance — All participants will receive a 8 lesson 3-month weight loss intervention. They will then be randomized. Those continuing with the intervention will receive 17 more lessons delivered face-to-face or via DVD over 15 months for a total of 18 months. Each lesson lasts approximately 1 hour and helps participants integrate healthy eating and physical activity into their lifestyles. Participants will also be encouraged to attend 13 community activities during the last 13 months of the intervention.
  Other Names: PILI 'Ohana Partnership
  Arms: DVD group; face-to-face group

SUMMARY:
This is a 5-year community-based participatory research intervention study with the goals of 1) conducting a more definitive study of weight loss maintenance in Native Hawaiians and Pacific Peoples and 2) identifying the aspects of the community-academic partnership that fosters a co-learning and co-equal environment.

DETAILED DESCRIPTION:
Obesity and overweight are well recognized public health concerns in the US and the magnitude of excess weight is greater among racial/ethnic minority populations. For NHs and PPs 70 to 80% of adults are estimated to be overweight or obese. Obesity-related disparities such as diabetes and heart disease (CVD) are also increasing among NHs and PPs. To address obesity and related disparities, a community-based participatory research (CBPR) partnership was formed entitled, the Partnership for Improving Lifestyle Interventions (PILI) 'Ohana Program (Pili meaning relationship and 'Ohana meaning family). The PILI 'Ohana Program (POP) consists of 5 community organizations and the Department of Native Hawaiian Health (DNHH) at the John A. Burns School of Medicine (JABSOM) of the University of Hawai'i (UH). With a 3-year CBPR planning grant from the National Center on Minority Health and Health Disparities (NCMHD), the POP was successful at establishing this community-academic partnership aimed at obesity-related disparities in Hawai'i and in implementing a pilot intervention to address weight loss maintenance (the PILI 'Ohana Intervention) in NHs and PPs, which serves as preliminary data for this application. The specific aims are as follow: 1) To identify the aspects of the PILI 'Ohana (family + community focused) Intervention deemed effective by former participants and community-peer educators of the pilot intervention. 2) To test whether a face-to-face or DVD delivery method of the PILI 'Ohana intervention is effective in improving weight loss maintenance versus a control group in NHs and PPs. 3) To identify the strengths of the PILI 'Ohana Program that supports a co-learning and co-equal environment.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Native Hawaiian, Filipino, or other Pacific Islander ethnic background;
* Age 18 years or older
* Overweight or Obese defined as BMI > 25 kg/m2 (NH or Pacific Islanders) or > 23 kg/m2 (Filipino ethnic background)
* Willing and able to follow a weight loss maintenance intervention program that could include 150 minutes of brisk walking per week (or equivalent) and a dietary regimen designed to maintain weight loss
* Able to identify at least one family, friend, or co-worker who would be willing to support the participant during the course of the study

Exclusion Criteria:

* Survival less than 6 months
* Planning to move out of the community during the intervention study period
* Pregnancy
* Any dietary or exercise restrictions that would prevent an individual from fully participating in the intervention protocol (i.e., end-stage renal disease on a renal diet, etc.)
* Any co-morbid condition (physical and mental disabilities) that would prevent the individual from participating in the intervention protocol (i.e., severe arthritis, hemi-paresis, major psychiatric illness, eating disorders, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | 18-months
  Amount of Weight loss in kilograms from baseline to 18 month follow-up

SECONDARY OUTCOMES:
Systolic/diastolic blood pressure | 18-months
  Systolic/diastolic blood pressure (mmHg) as measured by an electronic blood pressure device
Self-reported dietary fat intake | 18-months
  Self-reported dietary fat intake using an 18-item Food Frequency Questionnaire
Self-reported physical activity | 18-months
  Self-reported physical activity frequency and intensity using a 3-item brief physical activity questionnaire
Physical functioning | 18-month
  Physical functioning as measured by distance walked in feet via a 6-minunte Walk Test
Self-reported health beliefs | 18-month
  Self-reported health beliefs associated with diet, physical activity, and weight using a standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Kaholokula, PhD, Principal Investigator — University of Hawaii
Locations (4):
- United States (4):
  - Hawaii Maoli, Honolulu, Hawaii
  - Ke Ola Mamo, Honolulu, Hawaii
  - Kula no na Po'e Hawaii, Honolulu, Hawaii
  - Kokua Kalihi Valley, Honolulu, Hawaii

REFERENCES:
- [Derived] Sinclair KA, Zamora-Kapoor A, Townsend-Ing C, McElfish PA, Kaholokula JK. Implementation outcomes of a culturally adapted diabetes self-management education intervention for Native Hawaiians and Pacific islanders. BMC Public Health. 2020 Oct 20;20(1):1579. doi: 10.1186/s12889-020-09690-6. PMID 33081736
- [Derived] Sinclair KA, Makahi EK, Shea-Solatorio C, Yoshimura SR, Townsend CK, Kaholokula JK. Outcomes from a diabetes self-management intervention for Native Hawaiians and Pacific People: Partners in Care. Ann Behav Med. 2013 Feb;45(1):24-32. doi: 10.1007/s12160-012-9422-1. PMID 23086589